CLINICAL TRIAL: NCT06561074
Title: A Phase 2 Study to Evaluate Efficacy of Calaspargase Pegol-mknl and Decitabine Combined With Venetoclax in Pediatric, Adolescent, and Young Adult Patients With Relapsed/Refractory T-cell Acute Lymphoblastic Leukemia (T-ALL) and T- Cell Lymphoblastic Lymphoma (T-LLy)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0416; NCI-2024-06907 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-Cell Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Decitabine; venetoclax; calaspargase pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment w/Calaspargase pegol-mknl + Decitabine + Venetoclax (Experimental)
  Interventions: Drug: Decitabine; Drug: Venetoclax; Drug: Calaspargase pegol-mknl

INTERVENTIONS:
Drug: Decitabine — Given by vein
  Other Names: Dacogen
Drug: Venetoclax — Given by mouth
  Other Names: ABT-199, GDC-0199
Drug: Calaspargase pegol-mknl — Given by vein

SUMMARY:
To learn if giving the study drugs calaspargase pegol-mknl and decitabine in combination with venetoclax can help to control relapsed/refractory T-ALL and T-LLy. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives:

To characterize the clinical efficacy of Calaspargase pegol-mknl and Decitabine in combination with Venetoclax in pediatric, adolescent, and young adult patients with relapsed/refractory T-ALL/T-LLy based upon the complete response rate (CR).

Secondary Objectives:

To summarize efficacy per response rate, overall survival (OS), event free survival (EFS), and minimal residual disease (MRD) negativity rate.

To summarize the incidence, prevalence, and severity of adverse drug reactions according to common terminology criteria for adverse events (CTCAE) NCI CTCAE version 5.0.

• To summarize the effect of this treatment combination on patients transitioning to Hematopoietic stem cell transplant (HSCT) i.e., number and percentage of patients that are able to proceed to HSCT.

To evaluate calaspargase pegol-mknl pharmacokinetics in relapsed refractory patients and investigate its correlation with asparagine levels.

Exploratory Objectives:

To summarize associations between the genomic alterations in ALL (current biomarker expression of the disease) with relation to the incidence of proceeding to HSCT in patients with PR or stable disease (SD) after the induction cycle(s).

To evaluate the effect of anti-PEG and anti-ASP antibodies (PEG-ASP) on calaspargase enzyme levels, and effect of calaspargase pegol-mknl pharmacokinetics on toxicities and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric, adolescent, or young adult patients who have relapse or refractory T-cell lymphoblastic leukemia (T-ALL) or T-Cell lymphoblastic lymphoma (T-LLy) according to 2017 WHO classification and NCCN v1 2021.
2. Patients have adequate performance status (ECOG ≤2) for patients≥16 years old, Lansky score >50 for patients<16 years old.
3. Patients must be 1mo to 21 years of age at time of signing/or having proxy sign the informed consent.
4. Patients with asymptomatic CNS disease are eligible (see also Exclusion Criterion #2 in section 4.2.)
5. The following conditions are allowed on study: conditions requiring systemic glucocorticoid use, such as autoimmune disease, acute or chronic controlled graft versus host disease (GVHD) or severe asthma. Patients are also allowed up to 5 days of glucocorticoids as cytoreduction in combination with up to 3 doses of cyclophosphamide (200 mg/m2/day) are allowed as standard pre-phase treatment up to 1 day before start of study treatment or cytarabine up to 2gm/m2. This can also be discussed with PI.
6. Patients must have adequate organ function and laboratory results (obtained within 14 days of enrolment:

   1. Total serum bilirubin ≤1.5 x upper limit of normal (ULN). Patients with known Gilbert's syndrome may have a total bilirubin up to ≤3 x ULN.
   2. Adequate renal function (creatinine clearance ≥ 30 mL/min) unless related to disease.
   3. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤3 x ULN; ≤5 x ULN unless in case of suspected leukemic liver involvement
   4. Amylase, Lipase and Triglycerides must be WNL prior to administration of calaspargase pegol-mknl. If the lab values are outside the normal range, the treating physicians can discuss dosing/enrolling per PI discretion.
7. Females of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (β-HCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 3 months following the last dose of study drug. Effective methods of birth control include:

   1. Birth control pills, skin patches, birth control injections, implants (placed under the skin by a health care provider)
   2. Intrauterine devices (IUDs) and intra-uterine hormone-releasing systems (IUS)
   3. Condom
   4. Abstinence
   5. Bilateral tubal occlusion/ligation or Bilateral tubal occlusion/ligation by hysteroscopy with a hysterosalpingogram to confirm the procedure's success
8. Males need to inform the doctor right away if the partner becomes pregnant or suspects pregnancy. While in this study and for 90 days after the last treatment the patient should not donate sperm for the purposes of reproduction. He will need to use a condom while in this study and for 90 days after the last treatment.
9. Patients must have had at least 30 days between prior hematopoietic stem cell transplant and first dose of study drug.
10. Patients able and willing to swallow tablets or use oral dispersible tablets. No liquid formulation is available.

Exclusion Criteria:

1. Past or current history of a secondary or other primary tumor or a chronic myeloid leukemia (CML) blast crisis with exception of:

   uratively treated non-melanomatous skin cancer, other primary solid tumor treated with curative intent and no known active disease present, and no treatment administered during the last 2 years
2. Presence of clinically significant uncontrolled CNS pathology such as epilepsy, paresis, aphasia, stroke, severe brain injuries, organic brain syndrome, or psychosis.

   Presence of the following are allowed: headaches, vomiting, nerve palsy
3. Significant traumatic injury or major surgery (major surgery means opening of a body cavity, e.g., thoracotomy, laparotomy, laparoscopic organ resection, and major orthopedic procedures, e.g. joint replacement, open reduction, and internal fixation) within 14 days of scheduled dosing day 1.
4. Male or female subjects of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with institution's standards.
5. Patients with uncontrolled infections (viral, bacterial, or fungal) per PI's discretion. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
6. Medical history of cardiovascular disease such as:

   Clinically significant cardiac disease including congestive heart failure (NYHA class III or IV), arrhythmia or conduction abnormality requiring medication, or cardiomyopathy.
7. Female patient who is pregnant or breastfeeding. Female patient who is considering becoming pregnant during the study; or within approximately 30 days after the last dose of venetoclax, 3 months after the last dose of calaspargase or 6 months after the last dose of decitabine. For decitabine and calaspargase, also see the study drugs product label for pregnancy precautions. Male patient who is considering fathering a child within approximately 30 days or donating sperm during the study, within approximately 90 days after the last dose to venetoclax, calaspargase and decitabine. For all study drugs, also see the relevant chemotherapy product label for not fathering a child and donating sperm.
8. Patients may be excluded if they are currently enrolled in another ongoing clinical trial with investigational products
9. Liver cirrhosis or other active severe liver disease or with suspected active alcohol abuse.
10. Patients who are unable or unwilling to comply with all study requirements for clinical visits, examinations, tests, and procedures.
11. If patient has not recovered from grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy- (exception no grade 3 or higher peripheral neuropathy) from previous chemotherapy, surgery, radiation before the start of study drugs.
12. Pancreatitis: Patients will be excluded in the presence of Grade 3 or 4 pancreatitis or if history of anaphylaxis or grade 3 pancreatitis from asparaginase.
13. Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the Investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
14. History of serious hypersensitivity reactions including anaphylaxis to pegylated L-Asparaginase therapy.
15. Known history of coagulopathy (e.g., hemophilia and know protein S deficiency).
16. Active thromboembolic event(s) (i.e., symptomatic despite initiation of anti-coagulation therapy), or history of CNS thromboses.
17. Patients should not have received the following within 7days prior to the first dose of study drug: Strong and moderate CYP3A inducers.
18. Malabsorption syndrome or any other condition that precludes enteral administration.
19. Has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit or used a strong or moderate CYP3A inhibitor within 2 days prior to the first dose of venetoclax.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: David McCall, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org